CLINICAL TRIAL: NCT06465693
Title: Personalized Nutrition Therapy Using Continuous Glucose Monitoring to Improve Outcomes in Type 2 Diabetes Mellitus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MED-2023-32168
Record Dates: First submitted 2024-06-13; First posted 2024-06-20 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Nutrition Therapy

STUDY DESIGN:
Intervention Model Description: will compare CGM plus nutrition therapy to nutrition therapy only in participants with type 2 diabetes
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group1 (Experimental): After consent, screening, and a 10-day run-in period, eligible participants will be randomly assigned to unblinded CGM plus nutrition therapy
  Interventions: Device: Unblinded CGM plus nutrition therapy
- Group 2 (Active Comparator): After consent, screening, and a 10-day run-in period, eligible participants will be randomly assigned to nutrition therapy only
  Interventions: Behavioral: Nutrition therapy only

INTERVENTIONS:
Device: Unblinded CGM plus nutrition therapy — will receive evidence-based nutrition guidance by a certified and licensed registered dietitian (RD), including information on portion sizes, macronutrient types, and effect of carbohydrates on blood glucose.
  will receive Dexcom G6 Pro CGMs to wear throughout the study. The CGM will be unblinded so that the glucose data will be available in real time to the participant and investigators. The dietitian and participant will review CGM data together
  Arms: Group1
Behavioral: Nutrition therapy only — will receive evidence-based nutrition guidance by a certified and licensed registered dietitian (RD), including information on portion sizes, macronutrient types, and effect of carbohydrates on blood glucose.
  Arms: Group 2

SUMMARY:
Nutrition guidelines state that multiple eating patterns are effective for type 2 diabetes and that therapy should be individualized. Yet many nutrition plans fail to account for interpersonal variability in blood glucose response to meals. This diminishes the ability of dietary interventions to optimize glycemic control and may lessen patient satisfaction, self--efficacy, and adherence. Continuous glucose monitoring (CGM) can facilitate behavior change in type 2 diabetes and has been associated with improved outcomes in nutrition intervention studies; this literature is limited by small study sample sizes and heterogeneity of study design and outcomes, and more data are needed. CGM could be a powerful tool for adapting a nutrition plan based on blood glucose response at an individual level. This study will test the use of CGM to personalize nutrition therapy compared to nutrition therapy alone (without CGM) for participants with type 2 diabetes who are not meeting glycemic treatment goals.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Have a previous diagnosis of type 2 diabetes
* HbA1c of 7.0 - 9.5%
* Stable medications for diabetes for at least 3 months prior to enrollment, with no plans to change medications or doses during the intervention period.

Exclusion Criteria:

* Type 1 diabetes
* Treatment with insulin, sulfonylurea, or meglitinide
* Use of a nondiabetic medication affecting blood glucose (e.g. corticosteroid)
* BMI <25 kg/m2
* Weight change >5 pounds in the 3 months prior to enrollment
* Estimated glomerular filtration rate <60 ml/minute/1.73 m2
* Pregnant or breastfeeding
* Anemia (which affects HbA1c)
* Presence of any disease that would make adherence to the protocol difficult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
HgbA1c | week 12

SECONDARY OUTCOMES:
Glucose variability/coefficient of variation | week 12
  using CGM data
mean glucose | week 12
  using CGM data
time in range (glucose 70-180 mg/dl) | week 12
  using CGM data
time above range (glucose 70-180 mg/dl) | week 12
  using CGM data
Weight | week 12
Fasting plasma glucose | week 12
Fasting serum insulin | week 12
Serum lipid panel | week 12
Intervention Acceptability Questionnaire | week 12
Diabetes Treatment Satisfaction Questionnaire (DTSQ) | week 12
Diet Satisfaction Questionnaire (DSat-28) | week 12
Diabetes Management Self-Efficacy Scale (DMSES) | week 12
Medication Effect Score | week 12

CONTACTS AND LOCATIONS:
Overall Officials: Anne Bantle, MD,MS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States